CLINICAL TRIAL: NCT00376181
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled Study to Determine the Efficacy, Safety, and Tolerability of AD-4833-536 in the Treatment of Subjects With Type 2 Diabetes
Brief Title: Efficacy, Safety and Tolerability of Pioglitazone-Azilsartan in Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Combination formulation concerns
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-OPI536-003; U1111-1114-1098 (Registry Identifier: WHO)
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; hypertension; blood pressure; diastolic blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Pioglitazone; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pioglitazone 45 mg/Azilsartan 20 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and Azilsartan
- Pioglitazone 45 mg/Azilsartan 40 mg QD (Experimental)
  Interventions: Drug: Pioglitazone and Azilsartan
- Pioglitazone 45 mg QD (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone and Azilsartan — Pioglitazone 45 mg and Azilsartan 20 mg combination tablets, orally, once daily for up to 24 weeks.
  Other Names: Actos; AD-4833; TAK-536
  Arms: Pioglitazone 45 mg/Azilsartan 20 mg QD
Drug: Pioglitazone and Azilsartan — Pioglitazone 45 mg and Azilsartan 40 mg combination tablets, orally, once daily for up to 24 weeks.
  Other Names: Actos; AD-4833; TAK-536
  Arms: Pioglitazone 45 mg/Azilsartan 40 mg QD
Drug: Pioglitazone — Pioglitazone 45 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: Actos; AD-4833
  Arms: Pioglitazone 45 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pioglitazone-azilsartan, once daily (QD), in subjects with type 2 diabetes mellitus with poor glycemic control.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic disease. In the United States, an estimated 21 million people have diabetes, with type 2 diabetes occurring in 90% to 95% of cases. Hypertension (high blood pressure) affects approximately 50 million individuals in the United States. The association of diabetes and hypertension is increased in this population; hypertension is more common in persons with diabetes while individuals with hypertension are 2.5 times more likely to develop diabetes than those who have normal blood pressure. As a result, more than 70% of adults with diabetes have hypertension (defined as having blood pressure greater than or equal to 130/80 mm Hg or using prescription medication for hypertension).

Patients with type 2 diabetes and hypertension are at high risk of other illnesses and death. Diabetes and hypertension are associated with insulin resistance (normal amounts of insulin are no adequate to produce a normal insulin response from fat, muscle and liver cells). and hyperinsulinemia (excess levels of insulin in the blood), which are independent risk factors for cardiovascular (heart vessel) disease. Individuals with type 2 diabetes carry a 2 to 4- time greater risk of cardiovascular disease and stroke compared with the general population. Uncontrolled hypertension also is associated with an increased risk of cardiovascular disease and stroke.

Takeda Global Research and Development Center, Inc. is developing a fixed-dose combination product, AD-4833-536. AD-4833-536 is a combination of AD-4833 (pioglitazone) and TAK-536 (azilsartan). Pioglitazone is an oral antidiabetic agent that acts by reducing insulin resistance and approved for treatment of adult patients with type 2 diabetes mellitus. Azilsartan is a angiotensin II receptor blocker that modulates the renin-angiotensin-aldosterone system that regulates blood pressure.

ELIGIBILITY:
Inclusion Criteria

* Type 2 diabetes with glycosylated hemoglobin of greater than or equal to 9.0 to less than or equal to 11.0% at Screening.
* Documented hypertension.
* On a stable diet and exercise program in addition to metformin alone or combination of metformin and a sulfonylurea for a minimum of 8 weeks prior to screening.
* If receiving antihypertensive therapy, must be on no more than 3 agents and be on a stable regimen.
* Clinical laboratory evaluations (including clinical chemistry, hematology, and urinalysis) within the reference range unless the results are deemed not clinically significant for inclusion into this study by the investigator.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria

* Type 1 diabetes mellitus.
* Diastolic blood pressure greater than 104 mm Hg at randomization visit.
* Currently taking an angiotensin II-receptor blocker.
* Unstable angina or heart failure of any etiology with New York Heart Association functional class III or IV.
* History of myocardial infarction, cerebrovascular accident (stroke), percutaneous coronary intervention, coronary artery bypass graft or transient ischemic attack within the previous six months.
* Clinically significant cardiac conduction defects.
* Secondary hypertension of any etiology.
* Body mass index greater than 45 kg/m2
* Has significant renal dysfunction.
* History of drug abuse or a history of alcohol abuse within the past 2 years.
* Previous history of cancer, other than basal cell carcinoma or stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to the first dose of study drug.
* Alanine transaminase or aspartate transaminase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
* Serum potassium greater than the upper limit of normal.
* Currently participating in another investigational study or has participated in an investigational study within 30 days prior to Randomization.
* Any other serious disease or condition that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
* Is hypersensitive to angiotensin II receptor blockers.
* Is hypersensitive to thiazolidinediones.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * any anti-diabetic agent (including thiazolidinediones and/or insulin) except for metformin or a combination of metformin and a sulfonylurea
  * niacin more than 200mg per day
  * tricyclic antidepressants or phenothiazines
  * Angiotensin II receptor blockers
  * Thiazolidinediones
  * Insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin. | Baseline and Week 24
  The change between the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 or including final visit, and Glycosylated Hemoglobin collected at baseline.

SECONDARY OUTCOMES:
Change from Baseline in Diastolic Blood Pressure | Baseline and Weeks 4, 8, 12, 16, 20, and 24.
  The change between Diastolic Blood Pressure measured at each week indicated including final visit and Diastolic Blood Pressure measured at baseline.
Change from Baseline in Systolic Blood Pressure | Baseline and Weeks 4, 8, 12, 16, 20, and 24
  The change between Systolic Blood Pressure measured at each week indicated including final visit and Systolic Blood Pressure measured at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (73):
- United States (59):
  - Huntsville, Alabama
  - Tallassee, Alabama
  - Little Rock, Arkansas
  - Auburn, California
  - Bakersfield, California
  - Buena Park, California
  - Chula Vista, California
  - Huntington Park, California
  - Los Gatos, California
  - Norwalk, California
  - Orangevale, California
  - Sacramento, California
  - Stockton, California
  - Deerfield Beach, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Marianna, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Dunwoody, Georgia
  - Chicago, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Prince Frederick, Maryland
  - Livonia, Michigan
  - Saint Clair Shores, Michigan
  - Las Vegas, Nevada
  - Trenton, New Jersey
  - Albany, New York
  - Johnson City, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Buckingham, Pennsylvania
  - Jeannette, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - New Tazewell, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Euless, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McKinney, Texas
  - Midland, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Virginia Beach, Virginia
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Chile (2):
  - Santiago
  - Temuco
- Mexico (5):
  - León, Guanajuato
  - Zapopan, Jalisco
  - Monterrey, Nuevo León
  - Guadalajara
  - Mexico City
- Peru (4):
  - Arequipa
  - Lambayeque
  - Lima
  - Trujillo

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI